CLINICAL TRIAL: NCT00910078
Title: Serum Free Light Chain Ratio, Total Kappa/Lambda Ratio, and Immunofixation as Prognostic Factors in Multiple Myeloma.
Brief Title: Serum Free Light Change in Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Other Study IDs: sFLC r, KLR and IFIX
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Multiple Myeloma
Keywords: Total kappa and lambda ratio; Stem cell transplantation; Serum immunofixation
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to evaluate the predictive role of free Kappa/Lambda ration in Multiple Myeloma post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected with Multiple Myeloma who underwent autologous or auto/allogenic stem cell transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of patients undergoing autolog transplantatio
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera S. Giovanni Battista, Torino, Torino, Italy